CLINICAL TRIAL: NCT04770688
Title: Safety and Efficacy of Osimertinib Combined With Anlotinib in EGFRm+, Treatment-naïve IIIb/IV NSCLC Patients: a Prospective, Single Arm, Phase Ib/IIa Study
Brief Title: Advanced Lung Tumor Treated by Osimertinib Plus Anlotinib
Acronym: AUTOMAN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Professor, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-18-13979
Record Dates: First submitted 2021-02-09; First posted 2021-02-25 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Non-Small Cell Lung Cancer With EGFR Mutation; Locally Advanced Solid Tumor; Metastatic Cancer; Adenocarcinoma of Lung
MeSH Terms: conditions — Neoplasm Metastasis; Adenocarcinoma of Lung | interventions — osimertinib; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib + Anlotiib (Experimental): Escalating doses and expanding doses of Anlotinib administered with Osimertinib
  Interventions: Drug: Osimertinib; Drug: Anlotinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib, 80mg, QD, p.o.
  Other Names: Tagrisso
Drug: Anlotinib — (Phase Ib) Anlotinib, from 8mg to10mg to 12mg, QD, p.o. from day 1 to 14 of a 21-day cycle.
  (Phase IIa)Anlotinib, given at RP2D dose QD, p.o. from day 1 to 14 of a 21-day cycle.
  Other Names: Focus V

SUMMARY:
This is a prospective, single arm, phase Ib/IIa study. Up to 25 patients will be enrolled into the study (Part A: 2-18; Part B: 7-19). The study has been designed to allow an investigation of the optimal combination dose and schedule whilst of Osimertinib plus Anlotinib in patients with EGFRm+, treatment-naïve IIIb/IV Non-Small Cell Lung Cancer (NSCLC) ensuring the safety of patients with intensive safety monitoring. There are two main parts to this study; Part A, Combination dose finding and Parts B, Dose expansion.

DETAILED DESCRIPTION:
Part A has been designed to identify the recommended dose of the combination of Osimertinib plus Anlotinib for further clinical evaluation based upon assessment of the safety and tolerability data collected during the first 21 days (cycle 1, 21 days per cycle). A cycle of study treatment will be defined as 21 days. Dosing will begin at Osimertinib 80mg QD continuously and Anlotinib 8mg QD from day1 to 14 of a 21-day cycle. In the first 6 patients, a delay of at least 21 days (the first group of 3 patients) and a delay of at least 7 days (the second group of 3 patients) will be mandatory between the administration of the first dose to the first patient and administration of first dose to subsequent patients. Patients will be enrolled to ensure a minimum of 3 and a maximum of 6 evaluable patients per cohort. Dose escalation and de-escalation will follow the scheme below, according to the following logic：If no dose-limiting toxicity (DLT) is observed (for definition see Section 4.1.3) in a cohort of 3 evaluable patients then dose escalation may occur. Dose increases will be permitted after review of data from a minimum of 3 evaluable patients has been performed.

* If one patient experiences a DLT in a group of 3 evaluable patients then the cohort will be expanded to include 6 evaluable patients. If only one DLT is observed in the complete cohort of 6 evaluable patients then dose escalation may occur.
* If 2 or more patients experience a DLT in a group of up to 6 patients, irrespective of the number of patients enrolled, the dose will be considered not tolerated and recruitment to the cohort and dose escalation will cease.

Safety will be intensively monitored in part A. If RP2D was not reached in Part A, Part B would not be initiated. If RP2D was reached in Part A, eligible patients in part B will be enrolled and receive Osimertinib (80mg QD, continuously) plus Anlotinib (RP2D, QD from day 1 to 14 of a 21-day cycle) till disease progression (PD) or unacceptable toxicity, with the aim to further evaluate the safety, tolerability and efficacy in terms of ORR, DCR, DOR, PFS, overall survival at 12 months.

For all eligible patients (Part A and Part B), tissue and/or blood samples at baseline and PD will be collected to understand the resistance profile.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study subjects should fulfil the following criteria:

  1. Provision of informed consent prior to any study specific procedures.
  2. Aged at least 18 years.
  3. Histologically or cytologically confirmed locally advanced/metastasis NSCLC, adenocarcinoma of the lung (AJCC Eighth Edition TNM Stage ⅢB to stage Ⅳ), not amenable to curative surgery or radiotherapy.
  4. WHO/Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1 with no deterioration over the previous 2 weeks and a minimum life expectation of at least 12 weeks.
  5. The tumour harbours one of the most common EGFR mutations known to be associated with EGFR-TKI sensitivity (exon 19 deletion; L858R) either alone or in combination with other EGFR mutations as confirmed by a local test.
  6. No prior systemic anti-cancer, EGFR-TKI, or immunotherapy therapy for their locally advanced or metastasis disease (biopsy will be at time of diagnosis of locally advanced/metastasis disease).
  7. At least one lesion is measurable based on Response Evaluation Criteria in Solid Tumours (RECIST 1.1).
  8. Adequate bone marrow reserve and organ function as follows:
* Absolute neutrophils count (ANC) ≥1.5x109/L (band neutrophil and segmented neutrophil), platelets >100x109/L and Hb ≥90g/L.
* Hepatic: total bilirubin ≤1.5 times upper limit of normal (ULN).
* Alkaline phosphatase, alanine transaminase (ALT) and aspartate transaminase (AST)≤3.0 ULN (or ≤5 ULN in case of known liver involvement).
* Renal: Serum Creatinine ≤1.5ULN, creatinine clearance (CCr) ≥50mL/min 9. Female patients of childbearing potential must be using adequate contraceptive measures (see Restrictions, Section3.5), must not be breast feeding, and must have a negative pregnancy test prior of study treatments and confirmed prior to start of dosing on day 1. Otherwise, they must have evidence of non-childbearing potential as defined below:
* Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
* Women under 50 years would be consider post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
* Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation 10. Male patients must be willing to use barrier contraception, i.e., condoms (see Restrictions, Section 3.5) 11. Optional provision of an unstained, archived tumour tissue samples or fresh tissue and/or blood in a quantity sufficient to allow for central NGS testing (FFPE slices or fresh tumor tissue or blood at sufficient amount for NGS analysis).

Exclusion Criteria:

- Subjects must not enter the study if any of the following exclusion criteria are fulfilled:

1. Patients with non-lung adenocarcinoma including lung squamous carcinoma, or mixed histology, etc.
2. Treatment with any of the following:

   * Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   * Patients currently receiving (or unable to stop use prior to receiving the first dose of study drug) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3-week prior) (Appendix B). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
   * Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
3. Any concurrent and/or other active malignancy that has required treatment within 5 years of first dose of study drug.
4. Any unresolved toxicities from prior systemic therapy (e.g., adjuvant chemotherapy) greater than CTCAE grade 1 at the time of starting study drug with the exception of alopecia and grade 2, prior chemotherapy-induced neuropathy.
5. Spinal cord compression, symptomatic and unstable brain metastases, except for those patients who have completed definitive therapy, and have had a stable neurological status for at least 2 weeks after completion of definitive therapy. Patients may be on corticosteroids to control brain metastases if they have been on a stable dose for 2 weeks (14 days) prior to the start of study treatment and are clinically asymptomatic.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Recent active digestive disease such as duodenal ulcers, ulcerative colitis, ileus, ect., intestinal perforation, intestine fistula, or other conditions may lead to gastrointestinal bleeding or perforation which regimented at investigators' discretion.
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of Osimertinib and Anlotinib.
9. Cardiac function evaluation: LVEF <50%, a recent history of MI in 6 months, severe/unstable angina or coronary bypass surgery, or cardiac insufficiency ≥ NYHA 2. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, interval >250 msec.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN), congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
   * Past medical history of ILD, drug-induced ILD, radiation pneumonitis which require steroid treatment, or any evidence of clinically active ILD.
   * Previous allogenic bone marrow transplant.
   * Pregnant or lactating woman who are breast feeding.
   * A history of organ transplantation and long-term immunosuppressive medication.
   * History of hypersensitivity to active or inactive of Osimertinib or Anlotinib or drugs with a similar chemical structure or class to osimertinib or Anlotinib.
10. Judgment by the Investigator that the patients should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.; or other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II Dose(RP2D) | Up to approximately 6 months
  RP2D is defined as the dose cohort as follows: (1). If 2 or more of 6 patients in cohort 1 experienced a DLT, the combination would not be considered tolerable. There would be no RP2D and no dose expansion. (2). If none of the first 3 patients or 1 of 6 patients in starting dose cohort 1 experienced a DLT, dose escalation to cohort 2 would be done in the next 3 to 6 patients. If 2 or more patients experienced a DLT in up to 6 patients in cohort 2, the RP2D will defined as Osimertinib 80mg and Anlotinib 8mg. (3).If none of the first 3 patients or 1 of 6 patients in cohort 2 experienced a DLT, dose escalation to cohort 3 would be done in the next 3 to 6 patients. If 2 or more patients experience a DLT in up to 6 patients in cohort 3, the RP2D will defined as Osimertinib 80mg and Anlotinib 10mg. (4). If none of the first 3 patients or 1 out of 6 patients experienced a DLT in cohort 3, the RP2D would be Osimertinib 80mg and Anlotinib 12mg.
ORR according to RECIST Version 1.1 | Up to approximately 3 years following the first dose of study drug
  According to RECIST 1.1, the proportion of subjects whose tumors were assessed as CR+PR by subcenter imaging evaluation was recorded from the time they were first treated until disease progression or initiation of a new anticancer treatment.

SECONDARY OUTCOMES:
Dose-limiting toxicity (DLT) | occurs from the first dose of study drug (Day 1, Cycle 0) up to the last day of Cycle 1 (21 days after start of dosing)
  A DLT is defined as any toxicity not attributable to the disease or disease-related processed under investigation.
Disease Control Rate (DCR) | Up to approximately 3 years following the first dose of study drug
  Proportion of patients whose tumors shrink or remain stable for a certain period of time, including CR, PR, and SD;
Duration of disease remission (DOR) | Up to approximately 3 years following the first dose of study drug
  The time from objective tumor remission (CR or PR) to objective tumor progression or death for any reason (whichever occurs first) was recorded for the first time.
Disease progression-free survival(PFS) | Up to approximately 3 years following the first dose of study drug
  The time from the first use of the drug into the group to the progression of the disease or death (in terms of the first appearance)
Overall Survival(OS) | Up to approximately 5 years following the first dose of study drug
  The time from the first use of the drug into the group to the time of all-cause death. For the subjects who were still alive at the last follow-up, the OS was deleted according to the time of the last follow-up. For the subjects who lost the follow-up, their OS was counted as data deletion according to the last confirmed survival time before the loss of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seto T, Kato T, Nishio M, Goto K, Atagi S, Hosomi Y, Yamamoto N, Hida T, Maemondo M, Nakagawa K, Nagase S, Okamoto I, Yamanaka T, Tajima K, Harada R, Fukuoka M, Yamamoto N. Erlotinib alone or with bevacizumab as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harbouring EGFR mutations (JO25567): an open-label, randomised, multicentre, phase 2 study. Lancet Oncol. 2014 Oct;15(11):1236-44. doi: 10.1016/S1470-2045(14)70381-X. Epub 2014 Aug 27. PMID 25175099
- [Result] Ichihara E, Hotta K, Nogami N, Kuyama S, Kishino D, Fujii M, Kozuki T, Tabata M, Harada D, Chikamori K, Aoe K, Ueoka H, Hosokawa S, Bessho A, Hisamoto-Sato A, Kubo T, Oze I, Takigawa N, Tanimoto M, Kiura K. Phase II trial of gefitinib in combination with bevacizumab as first-line therapy for advanced non-small cell lung cancer with activating EGFR gene mutations: the Okayama Lung Cancer Study Group Trial 1001. J Thorac Oncol. 2015 Mar;10(3):486-91. doi: 10.1097/JTO.0000000000000434. PMID 25695221
- [Result] Rosell R, Dafni U, Felip E, Curioni-Fontecedro A, Gautschi O, Peters S, Massuti B, Palmero R, Aix SP, Carcereny E, Fruh M, Pless M, Popat S, Kotsakis A, Cuffe S, Bidoli P, Favaretto A, Froesch P, Reguart N, Puente J, Coate L, Barlesi F, Rauch D, Thomas M, Camps C, Gomez-Codina J, Majem M, Porta R, Shah R, Hanrahan E, Kammler R, Ruepp B, Rabaglio M, Kassapian M, Karachaliou N, Tam R, Shames DS, Molina-Vila MA, Stahel RA; BELIEF collaborative group. Erlotinib and bevacizumab in patients with advanced non-small-cell lung cancer and activating EGFR mutations (BELIEF): an international, multicentre, single-arm, phase 2 trial. Lancet Respir Med. 2017 May;5(5):435-444. doi: 10.1016/S2213-2600(17)30129-7. Epub 2017 Apr 10. PMID 28408243
- [Result] Ninomiya T, Nogami N, Kozuki T, Harada D, Kubo T, Ohashi K, Kuyama S, Kudo K, Bessho A, Fukamatsu N, Fujimoto N, Aoe K, Shibayama T, Sugimoto K, Takigawa N, Hotta K, Kiura K. A phase I trial of afatinib and bevacizumab in chemo-naive patients with advanced non-small-cell lung cancer harboring EGFR mutations: Okayama Lung Cancer Study Group Trial 1404. Lung Cancer. 2018 Jan;115:103-108. doi: 10.1016/j.lungcan.2017.11.025. Epub 2017 Nov 28. PMID 29290249
- [Result] Porta R, Sanchez-Torres JM, Paz-Ares L, Massuti B, Reguart N, Mayo C, Lianes P, Queralt C, Guillem V, Salinas P, Catot S, Isla D, Pradas A, Gurpide A, de Castro J, Polo E, Puig T, Taron M, Colomer R, Rosell R. Brain metastases from lung cancer responding to erlotinib: the importance of EGFR mutation. Eur Respir J. 2011 Mar;37(3):624-31. doi: 10.1183/09031936.00195609. Epub 2010 Jul 1. PMID 20595147
- [Result] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Result] Han B, Li K, Zhao Y, Li B, Cheng Y, Zhou J, Lu Y, Shi Y, Wang Z, Jiang L, Luo Y, Zhang Y, Huang C, Li Q, Wu G. Anlotinib as a third-line therapy in patients with refractory advanced non-small-cell lung cancer: a multicentre, randomised phase II trial (ALTER0302). Br J Cancer. 2018 Mar 6;118(5):654-661. doi: 10.1038/bjc.2017.478. Epub 2018 Feb 13. PMID 29438373
- [Result] Becker A, Crombag L, Heideman DA, Thunnissen FB, van Wijk AW, Postmus PE, Smit EF. Retreatment with erlotinib: Regain of TKI sensitivity following a drug holiday for patients with NSCLC who initially responded to EGFR-TKI treatment. Eur J Cancer. 2011 Nov;47(17):2603-6. doi: 10.1016/j.ejca.2011.06.046. Epub 2011 Jul 23. PMID 21784628